CLINICAL TRIAL: NCT06131307
Title: The Effect of Paternalistic Leadership Training Given to Health Managers on Nurses' Motivation, Organizational Commitment, and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KSBUHSU52
Record Dates: First submitted 2023-11-02; First posted 2023-11-14 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-10

CONDITIONS: Paternalism; Motivation; Organizational Behavior
Keywords: Paternalistic leadership; Organizational commitment; Employee Performance; Nurses
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Managers of this group will be given paternalistic leadership training. Before the training, paternalistic leadership perception, motivation, organizational commitment, and performance levels will be measured. Two months after the paternalistic leadership training given to managers, the paternalistic leadership perception, motivation, organizational commitment and performance levels of the same participants will be measured again.
  Interventions: Procedure: Education
- Control group (No Intervention): Managers of this group will not be given paternalistic leadership training. At the same time as the first group, paternalistic leadership perception, motivation, organizational commitment, and performance levels will be measured.

INTERVENTIONS:
Procedure: Education — Paternalistic leadership training will be given to clinical manager nurses.
  Arms: Experimental group

SUMMARY:
Research on leadership behaviors has been ongoing since the early 1900s. As a result of these studies, many leadership types (charismatic, transformational, transactional, paternalist, etc.) have been defined according to the behaviors of leaders. In this research, the effect of paternalistic leadership on motivation, organizational commitment, and performance will be discussed. A paternalist leader is defined as a leader who has a virtuous and moral character, attaches importance to hierarchy, creates a family atmosphere in the workplace, knows his employees closely, stands by them in good and bad times, protects them like a father, and expects respect and loyalty from his employees in return for what he does.

The success of managers depends on their ability to motivate their subordinates to behave in a way that achieves organizational goals and on employees' use of their knowledge, abilities, and energy in this The success of an organization depends not only on how it develops the talents of its employees to the highest level but also on how it encourages its employees to commit to the organization's direction. For these reasons, motivation is an important issue for managers. The ability of organizations to operate effectively and efficiently and ensure their sustainability largely depends on the performance of their human resources.

In the studies carried out to date, the effect of paternalistic leadership on employee performance, work motivation, and organizational commitment has been examined, but there is no study investigating the effect of paternalistic leadership on nurses' motivation, organizational commitment, and performance after paternalistic leadership training is given to healthcare managers. Therefore, it is thought that this study will make a significant contribution to both healthcare managers and the literature. The aim of this research is to determine whether paternalistic leadership training given to healthcare managers has an effect on the motivation, organizational commitment, and performance of healthcare professionals.

DETAILED DESCRIPTION:
Research on leadership behaviors has been ongoing since the early 1900s. As a result of these studies, many leadership types (charismatic, transformational, transactional, paternalist, etc.) have been defined according to the behaviors of leaders. In this research, the effect of paternalistic leadership on motivation, organizational commitment, and performance will be discussed. A paternalist leader is defined as a leader who has a virtuous and moral character, attaches importance to hierarchy, creates a family atmosphere in the workplace, knows his employees closely, stands by them in good and bad times, protects them like a father, and expects respect and loyalty from his employees in return for what he does.

The success of managers depends on their ability to motivate their subordinates to behave in a way that achieves organizational goals and on employees' use of their knowledge, abilities, and energy in this The success of an organization depends not only on how it develops the talents of its employees to the highest level but also on how it encourages its employees to commit to the organization's direction. For these reasons, motivation is an important issue for managers. The ability of organizations to operate effectively and efficiently and ensure their sustainability largely depends on the performance of their human resources.

In the studies carried out to date, the effect of paternalistic leadership on employee performance, work motivation, and organizational commitment has been examined, but there is no study investigating the effect of paternalistic leadership on nurses' motivation, organizational commitment, and performance after paternalistic leadership training is given to healthcare managers. Therefore, it is thought that this study will make a significant contribution to both healthcare managers and the literature. The aim of this research is to determine whether paternalistic leadership training given to healthcare managers has an effect on the motivation, organizational commitment, and performance of healthcare professionals.

In order to prevent bias, patients will be included in the study groups according to the assignment made by the Randomizer.org program. Since the data will be transferred to the SPSS program and the analysis will be done by an independent statistician, the bias will also be controlled in the data evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Speaking Turkish,
* Working as a nurse for at least one year,
* No mental health problems

Exclusion Criteria:

* Being under 18 years of age,
* Not being able to speak Turkish,
* Working as a nurse for less than one year,
* Having a mental health problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Paternalistic leadership, motivation, organizational commitment, performans Scale | It is expected that the behavioral change will not change within two months.
  In the group that did not receive training (n = 90), a difference of 3 or more is not expected in the paternalistic leadership, motivation, organizational commitment and performance scale mean scores between the first and last measurements (two months).

SECONDARY OUTCOMES:
Paternalistic leadership, motivation, organizational commitment, performans Scale | The behavioral change is expected to occur within two months.
  204 / 5.000 Çeviri sonuçları Çeviri sonucu In the trained group (n=90), it is expected that there will be an increase of 3 or more in the paternalistic leadership, motivation, organizational commitment and performance scale average scores between the first and last measurements (two months).

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya health science univercity, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided